

Exit Interview- Chalo! 2.0 for increasing HIV testing and care engagement for MSM on the Internet

#### **Informed Consent Form**

## 1) Background of the study:

The Humsafar Trust is an LGBTQ-community based organization working in the field of LGBTQ health and rights for over 20 years. Chalo! 2.0 study is being conducted by the Humsafar Trust with an aim to use virtual platforms like WhatsApp to promote the health of men who like other men. We are asking you to participate in this interview since you have been with Chalo! 2.0 for 18 months as a study participant, and have contributed to the project and science by filling our survey. Through this interview, we want to understand your motivation to participate in the study, your engagement with the WhatsApp content and any services you accessed as part of the project. We are also interested to know any challenges or barriers you faced during your participation in Chalo! 2.0. It will be great to receive any recommendations or suggestions regarding making the process better.

## 2) What will happen during the study:

If you agree to participate, you will participate in a 30-45 minute interview. During the interview, a trained investigator will ask you questions about your motivation to participate in the study, your engagement with the WhatsApp content, any services you accessed as part of the project and any challenges or barriers you faced during your participation in Chalo! 2.0. This interview will take place either in person or over an internet-/voice-based platform such as a regular or a Skype/Whatsapp call/ Gmeet/Zoom and be audio-recorded and later transcribed for analyses. Please note that the interview is entirely confidential and all (if any) personal identifiers will be removed from the final transcript. Your answers and views will not be attributed to you in any way in our report and/or any of the publications and will not affect any of the services you seek at Humsafar. The audio-files will be destroyed a year after data collection and the other data after five years.

## 3) Possible Risks, Side Effects, and Discomforts:

This interview poses minimal quantifiable harm to your physical or mental well-being and has been designed as an extremely low risk activity. However, there is a risk of discomfort in that you may find some of the questions sensitive or personal. You can skip any questions you do not wish to answer or ask to end the interview at any point. You could also choose to withdraw consent mid interview following which your audio recording will be deleted.

#### 4) Possible Benefits:

There are no direct benefits to you for participating in this study, but the results of this work could improve our understanding of challenges at the participant level and inform to strengthening these processes for future scale up.



IRB APPROVAL DATE: 06/26/2024 IRB EXPIRATION DATE: 10/24/2024

5) Compensation paid to the research participants:

You will receive Rs.500 as an honorarium for your participation. The honorarium will be transferred to you via gpay or other e-money platforms once the interview concludes. Please note that this compensation will only be provided once and if the interview has concluded and indicated as closed by the interviewer.

# 6) Whom to call if any questions/problems/adverse event:

You waive no legal or health rights by participating in this research study. The Institutional Review Board (IRB) of the Humsafar Trust (India) and Albert Einstein College of Medicine (USA) has approved this research study. If you have questions about your rights as a research participant, you may contact the IRB Coordinator Ganesh Acharya who can notify the Site Principal Investigator – Ms. Shruta Rawat or the IRB Chairperson or the Albert Einstein College of Medicine, on the information below:

Ganesh Acharya, The Humsafar Trust, 3rd floor, Manthan Plaza, Nehru Road, Vakola, Santacruz (East), Mumbai – 400 055; Tel: 022-26673800]. You may also contact the IRB Chairperson, Dr. Chitra Nayak, by contacting the IRB Coordinator, Ganesh Acharya, at the contact number listed above or on hst.irb@humsafar.org.

The following are the details for the Einstein IRB: Albert Einstein College of Medicine, 1300 Morris Park Ave., Belfer Bldg #1002, Bronx, New York 10461. If you have questions regarding your rights as a research subject, you may contact the IRB office at +1-718-430-2253.

| You can print or sav can email you a copy | the this page if you wish to for your records. You can also contact us and we yof this form. |
|---|---|
| | CONSENT OF RESEARCH PARTICIPANT |
| I voluntarily give co | ox below, I indicate that I understand the language and study procedures and onsent to participate in this study. Further, I have been fully explained the guage I understand and consent to the same |

The Humsafar Trust Institutional Review Board

IRB NUMBER: 2018-9471
Abort Einstein College of Medicine IRB APPROVAL DATE: 06

IRB APPROVAL DATE: 06/26/2024 IRB EXPIRATION DATE: 10/24/2024

| I agree to participate |
|------------------------|
| Date: |
| Place: |